CLINICAL TRIAL: NCT04354337
Title: Sleep Innovations for Preschoolers With Arthritis (SIPA): Developing and Testing the Usability and Feasibility of a Self-Management Intervention
Brief Title: Sleep Innovations for Preschoolers With Arthritis (SIPA): Developing and Pilot Testing of a Self-Management Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Weichao Yuwen, Assistant Professor, School of Nursing, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008492; P30NR016585 (NIH)
Record Dates: First submitted 2020-03-10; First posted 2020-04-21 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Sleep deficiency; Self-management; Chronic disease
MeSH Terms: conditions — Arthritis, Juvenile; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): 8-weeks online program with weekly modules for parents to learn about specific sleep topics and implement behavioral changes to improve their child's sleep.
  Interventions: Behavioral: Sleep Innovations for Preschoolers with Arthritis (SIPA)

INTERVENTIONS:
Behavioral: Sleep Innovations for Preschoolers with Arthritis (SIPA) — The SIPA intervention is interactive and personalized. Every week, parent will receive an email sent automatically through the system with instructions for this week's activity, designed to take about 30 minutes to complete. The SIPA weekly modules will begin with a learning module, then direct participants through goal setting, anticipated barriers, and problem solving. The intervention site will include fillable responses to queries, instructions, and assignments. Tasks for parents and their young children will use multimedia elements to enhance delivery of information, such as links to videos and pictures targeting self-efficacy, motivation, and patient activation. Submissions and progress will be monitored by the study team, who will send email, call or text with reminders (whichever the family prefers) and answer questions as needed, review progress, and help problem solve any technology issues or barriers to implementing skills.

SUMMARY:
Behavioral sleep problems such as sleep onset delays and frequent night wakings are common among young children (2-5 years). Children with a chronic health condition such as juvenile idiopathic arthritis (JIA) are even more prone to sleep problems, which are also associated with disease-related symptoms such as pain and fatigue. Early childhood is a critical period for establishing healthy sleep habits and self-regulation skills and is therefore an opportune time to identify and address unhealthy sleep habits. The Sleep Innovation for Preschoolers with Arthritis (SIPA) project will develop and pilot test a technology-based sleep intervention for parents of young children with JIA.

DETAILED DESCRIPTION:
The SIPA study aims to develop and test the usability, feasibility, acceptability, and preliminary effectiveness of a technology-based sleep intervention - Sleep Innovation for Preschoolers with Arthritis (SIPA) - that provides JIA parents with the necessary tools (self-efficacy, motivation, activation) to set goals, problem solve, and improve sleep in young children with JIA. SIPA will address the causes of sleep deficiency including behavioral sleep problems (e.g., sleep onset delay, frequent night awakenings, and sleep onset association disorder) in preschoolers with JIA using a single-arm pre- and post-test pilot study. Investigators will pilot test the intervention with 18 parents and preschoolers with JIA. Investigators will assess the feasibility and acceptability of the intervention among users, as will as analyze its preliminary effectiveness in terms of changes in behavioral sleep problems in the preschoolers pre- and post-intervention. The specific aims are to:

Aim 1. Apply a user-centered iterative design approach to develop and test the usability of a technology- based sleep self-management intervention - Sleep Innovation for Preschoolers with Arthritis (SIPA) - for 2-5-year-old children (preschoolers) with juvenile idiopathic arthritis (JIA).

2. Describe the feasibility, acceptability, and preliminary effectiveness of the SIPA intervention to address the causes of behavioral sleep problems (e.g., frequent night awakenings, and sleep onset association disorder) that are the main cause of sleep deficiency in preschoolers with JIA using a single-arm pre- and post-test pilot study.

ELIGIBILITY:
Inclusion Criteria for children:

* diagnosed with JIA
* 2-to-5 years
* parent report of sleep problems or sleep less than 9 hours/day

Inclusion Criteria for parents:

* >18 years
* able to read/speak English

Exclusion Criteria for children:

* diagnosed primary sleep disorder (e.g., obstructive sleep apnea)
* positive screen on the Pediatric Sleep Questionnaire (> 0.33) for sleep-disordered breathing (investigators will suggest follow up with the child's primary care provider because treatment of this condition is beyond the scope this intervention)
* developmental delay
* co-morbid condition (asthma, diabetes)

Exclusion Criteria for parents:

* nightshift work that would interfere with performing bedtime activities with children
* diagnosed with a chronic illness that would interfere with completing study procedures
* lack of daily access to the Internet or mobile device

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-03-20 (Actual); Study Completion 2021-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Weichao Yuwen, PhD, RN, Principal Investigator — University of Washington- Tacoma
Locations (1):
- University of washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SIPA Website — https://depts.washington.edu/sipa/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment happened from 2020.5.1 - 2020.11.12 at a local medical clinic
Pre-assignment Details: The numbers are parent-child dyads, each dyad consist of one parent and one child.
Period: Overall Study
Arm/Group | Intervention Group
Started | 16 (16 dyads, 16 parents and 16 children)
Completed | 12 (12 Dyads, 12 parents and 12 children)
Not Completed | 4

BASELINE CHARACTERISTICS:
Population: 16 children; because this intervention is intended to improve children's sleep outcomes, we only collected demographic information about the children.
Arm/Group | Intervention Group
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 16 completed the demographic survey
  years | 3.6 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 16/16
  Participants
    Female | 12
    Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 16 completed the demographic survey
  Participants
    Hispanic or Latino | 1
    Not Hispanic or Latino | 15
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 16 completed the demographic survey
  Participants
    American Indian or Alaska Native | 2
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 1
    Black or African American | 0
    White | 11
    More than one race | 2
    Unknown or Not Reported | 0
Children's Sleep Habits Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Children's Sleep Habits Questionnaire (CSHQ) is a survey that assesses a child's sleep quality and quantity by asking parents to report on their child's sleep habits. The CSHQ has 45 items, including 33 scored questions and seven additional items. Parents rate each scored question on a three-point scale: usually, sometimes, and rarely. The total Sleep Disturbances score is calculated by adding up all the scored questions. All responses are totaled to create a Total Sleep Disturbance index (range from 33-99), with a score exceeding 41 suggesting the presence of a pediatric sleep disorder. Population: 16 completed
  units on a scale | 48.36 (8.05)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by Adherence
Description: Adherence is calculated by the total number of dyads completing all intervention modules divided by the total number of dyads enrolled.
Time Frame: immediately after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group
Number analyzed (Participants) | 16
Participants | 12

2. Primary Outcome: Children's Sleep Habits Questionnaire
Description: The Children's Sleep Habits Questionnaire (CSHQ) is a survey that assesses a child's sleep quality and quantity by asking parents to report on their child's sleep habits. The CSHQ has 45 items, including 33 scored questions and seven additional items. Parents rate each scored question on a three-point scale: usually, sometimes, and rarely. The total Sleep Disturbances score is calculated by adding up all the scored questions. All responses are totaled to create a Total Sleep Disturbance index (range from 33-99), with a score exceeding 41 suggesting the presence of a pediatric sleep disorder.
Time Frame: baseline; 8 weeks (immediately after intervention); and 3 months (study completion).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group
Number analyzed (Participants) | 12
score on a scale
  baseline | 48.36 (8.05)
  8 weeks | 40.82 (5.53)
  3 months | 38.90 (2.81)

ADVERSE EVENTS:
Time Frame: 10 months
Description: for child only; adverse event for parents were not collected.
Arm/Group | Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT04354337/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT04354337/ICF_001.pdf